CLINICAL TRIAL: NCT01875224
Title: Open-Label, Randomized Comparison of NODAT in Renal Transplant Patients Receiving a Nulojix (Belatacept) Regimen Versus Standard Therapy Immunosuppression
Brief Title: Comparison of NODAT in Kidney Transplant Patients Receiving Belatacept Versus Standard Immunosuppression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Bruce Kaplan, Chief of Abdominal Transplantation, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IM103-303
Record Dates: First submitted 2013-05-29; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: New Onset Diabetes After Transplant; Kidney Transplantation
Keywords: kidney transplant; diabetes after transplant; belatacept
MeSH Terms: interventions — Abatacept; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belatacept and CellCept (Experimental): Belatacept administered based on patient's weight once a month after initial period, Cellcept taken twice daily.
  Interventions: Drug: Belatacept
- Tacrolimus and CellCept (Active Comparator): Tacrolimus and CellCept taken twice daily based on patient response.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Belatacept
  Other Names: Nulojix
  Arms: Belatacept and CellCept
Drug: Tacrolimus — Standard administration of tacrolimus
  Other Names: Prograf
  Arms: Tacrolimus and CellCept

SUMMARY:
This study is being conducted to determine if belatacept is an appropriate alternative immunosuppressive medication (reducing the immune system's effect) when a kidney transplant patient develops new onset diabetes after transplant (NODAT). Patients who are diagnosed with NODAT will be approached with the opportunity to participate in this study. If they agree to participate, they will be randomized one-to-one (like a coin flip) to the study arm (belatacept) or the control arm (their current medication regimen). If a patient is randomized to the study arm, they will be tapered off of their current regimen when they have started receiving their monthly belatacept infusions. The control arm will mean the patient will continue their current, standard of care medications, but following the tacrolimus trough levels indicated within the study protocol. Different laboratory tests (i.e. fasting blood glucose) will be measured during the study to monitor the progression of NODAT in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be given by patient.
* Adult patients between age 18 and 65
* Thymoglobulin induction at the time of transplant
* Patient must be Epstein-Barr Virus seropositive

Exclusion Criteria:

* Patient who received an blood type incompatible transplant, or with T-cell or B-cell positive crossmatch
* Patients with Hepatitis B, Hepatitis C, HIV or a clinically significant systemic infection within 30 days prior to transplant
* History of stroke, severe cardiac disease or cardiac failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Increased insulin sensitivity | 12 months
  Increase in insulin sensitivity (HOMA-S) as calculated below:
  FIRI = fasting plasma insulin level
  FPG = fasting plasma glucose level
  HOMA-S (insulin sensitivity) is calculated as 22.5 / (FIRI * FPG)
Decreased insulin resistance | 12 months
  Decreased insulin resistance (HOMA-IR) as measured below:
  FIRI = fasting plasma insulin level
  FPG = fasting plasma glucose level
  HOMA IR (insulin resistance) is calculated as (FIRI * FPG) / 22.5

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kaplan, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States